CLINICAL TRIAL: NCT07393230
Title: Evaluation of the Effect of Bilateral Balanced Orbital Decompression on Orbital, Retinal, and Choroidal Macro and Microvascular Blood Flow Parameters in Thyroid-Associated Orbitopathy
Brief Title: Changes in Orbital Macrovascular and Intraocular Microvascular Blood Flow After Orbital Decompression Surgery in Patients With Thyroid Eye Disease
Acronym: BOD-VASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Burçin Göğüş Çamlı, Ophthalmologist, Department of Ophthalmology, Marmara University School of Medicine, Marmara University Pendik Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2023.423; 09.2023.423 (Registry Identifier: Marmara University School of Medicine Ethics Committee)
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thyroid Associated Orbitopathy
Keywords: Thyroid-Associated Orbitopathy; Balanced Orbital Decompression; Orbital Blood Flow; Retinal and Choroidal Microcirculation; OCT Angiography; Doppler Ultrasonography

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, interventional study in which patients with inactive thyroid-associated orbitopathy undergo balanced orbital decompression surgery. Clinical, orbital macrovascular, and retinal-choroidal microvascular parameters are evaluated before surgery and at predefined postoperative follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balanced Orbital Decompression Surgery (Experimental): Participants in this arm undergo balanced orbital decompression surgery performed for inactive thyroid-associated orbitopathy, with preoperative and postoperative clinical and vascular assessments.
  Interventions: Procedure: Balanced Orbital Decompression Surgery

INTERVENTIONS:
Procedure: Balanced Orbital Decompression Surgery — Balanced orbital decompression is performed under general anesthesia using a combined medial and lateral orbital wall approach with orbital fat removal, aiming to reduce orbital pressure and improve orbital and ocular circulation in patients with inactive thyroid-associated orbitopathy.
  Other Names: Combined medial and lateral orbital wall decompression with orbital fat excision

SUMMARY:
This study aims to evaluate the effects of balanced orbital decompression surgery in patients with inactive thyroid-associated orbitopathy. The study examines how the surgery influences blood flow in the orbit and microcirculation in the retina and choroid over time. Clinical findings, imaging results, and vascular changes before and after surgery will be analyzed to better understand the anatomical and functional outcomes of the procedure.

DETAILED DESCRIPTION:
Thyroid-associated orbitopathy (TAO) is an autoimmune condition that can lead to increased orbital tissue volume, proptosis, elevated intraocular pressure, and impaired venous outflow. In the inactive phase of the disease, balanced orbital decompression (BOD) is commonly performed to relieve orbital pressure and improve both anatomical and functional outcomes.

While the clinical benefits of orbital decompression are well established, its effects on orbital blood flow and intraocular microcirculation have not been sufficiently investigated, particularly over time. This study is designed to prospectively evaluate the impact of BOD on orbital macrovascular structures and retinal-choroidal microvascular networks in patients with inactive TAO.

Patients undergoing BOD for severe proptosis will be evaluated before surgery and at multiple postoperative follow-up visits. Assessments include clinical ophthalmologic examinations, intraocular pressure measurements, and imaging-based evaluation of orbital and intraocular circulation. Orbital macrovascular parameters will be assessed using Doppler ultrasonography, while retinal and choroidal microcirculation will be analyzed using optical coherence tomography angiography (OCTA).

The study aims to characterize time-dependent vascular changes following surgery and to explore the relationship between macrovascular and microvascular responses. By providing longitudinal data, this study seeks to improve understanding of how orbital decompression influences ocular perfusion and vascular regulation, contributing to a more comprehensive evaluation of surgical outcomes in inactive TAO.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of inactive thyroid-associated orbitopathy
* Presence of moderate-to-severe proptosis with indication for surgical orbital decompression
* Planned to undergo balanced orbital decompression surgery
* Ability to provide written informed consent
* Adequate image quality for OCTA and Doppler ultrasonography assessments

Exclusion Criteria:

* Active phase thyroid-associated orbitopathy
* Thyroid dysfunction or systemic condition contraindicating general anesthesia
* Proptosis due to causes other than TAO
* History of orbital radiotherapy
* Previous orbital or intraocular surgery
* Presence of retinal or choroidal pathology affecting vascular measurements
* History of systemic vasculitis or other vascular diseases
* Diabetes mellitus or systemic hypertension
* Use of systemic immunosuppressive therapy
* Age under 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Change in ophthalmic artery flow velocities | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in peak systolic velocity and end-diastolic velocity of the ophthalmic artery, measured in cm/s, assessed by color Doppler ultrasonography before and after surgery.
Change in central retinal artery flow velocities | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in peak systolic velocity and end-diastolic velocity of the central retinal artery, measured in cm/s, assessed by color Doppler ultrasonography before and after surgery.
Change in superior ophthalmic vein diameter | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in superior ophthalmic vein diameter, measured in millimeters (mm), assessed by magnetic resonance imaging before and after surgery.

SECONDARY OUTCOMES:
Change in superficial capillary plexus vessel density | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in vessel density of the superficial capillary plexus, expressed as a percentage (%), assessed by optical coherence tomography angiography before and after surgery.
Change in deep capillary plexus vessel density | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in vessel density of the deep capillary plexus, expressed as a percentage (%), assessed by optical coherence tomography angiography before and after surgery.
Change in choriocapillaris vessel density | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in vessel density of the choriocapillaris, expressed as a percentage (%), assessed by optical coherence tomography angiography before and after surgery.
Change in choroidal vascularity index | Baseline and postoperative follow-up visits at 1, 3, and 6 months
  Change in choroidal vascularity index (unitless), assessed by optical coherence tomography before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Department of Ophthalmology, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No